CLINICAL TRIAL: NCT02547090
Title: The Effect of Two Surgeons on Blood Loss and Operative Time in Cerebral Palsy (CP) Patients Undergoing Posterior Spinal Fusion
Brief Title: Minimizing Complications in Scoliosis Surgery in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 11-124
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CP who underwent PSF by two attendings in 2012
  Interventions: Procedure: The use of two attending surgeons during posterior spinal fusion
- CP who underwent PSF by a single surgeon from 2008-2010

INTERVENTIONS:
Procedure: The use of two attending surgeons during posterior spinal fusion — Patients in the experimental group received posterior spinal fusion with two attending surgeons. Patients in the control group received posterior spinal fusion with one attending surgeon and one first assist, which could be a resident, PA, or nurse.
  Groups: CP who underwent PSF by two attendings in 2012

SUMMARY:
Background:

Posterior spinal fusion (PSF) in children with cerebral palsy (CP) carries a high risk of complications and mortality. Complication rates have been reported as high as 45%, and infection rates typically reported at 15%. Efforts to improve efficiency by reducing operative time and blood loss could decrease these risks. The purpose of this study is to investigate the impact of utilizing two attending surgeons on blood loss, operative time, and complications in this population.

Methods:

This is a prospective, matched cohort analysis with a consecutive series of patients with CP who underwent PSF, with two attending surgeons, in 2012. These are matched with a control group that had a single-surgeon team (operative dates 2008-2010), assisted by a resident, PA, or RN-FA. The groups are compared using paired Student T-tests and chi square tests (significance set a p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy
* neuromuscular scoliosis requiring posterior spinal fusion (>50 degree Cobb)
* PSF from 2008-2012 at Phoenix Children's Hospital
* GMFCS IV or V

Exclusion Criteria:

* Diagnosis other than CP
* GMFCS I-III
* Previous spine deformity surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study group consisted of 25 consecutive patients with CP and progressive neuromuscular scoliosis who underwent PSF in 2012 with the use of a two surgeon team. The control group consisted of a consecutive series of patients with CP who underwent PSF by a single surgeon from 2008-2010 at the same institution. The control group was a cohort of patients matched for age, gender, weight and Cobb angle.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Complications due to PFS surgery | Post-operative hospital stay (up to 12 days)

SECONDARY OUTCOMES:
Surgical time | intraoperative
Estimated blood loss | intraoperative
Length of Stay | During hospitalization (up to 12 days)